CLINICAL TRIAL: NCT05650047
Title: Home OCT Guided Management Study of Subjects Diagnosed With Neovascular-AMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2022.004
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-12

CONDITIONS: Retinal Neovascularization
Keywords: AMD self-scanning Home-OCT
MeSH Terms: conditions — Retinal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the last 25 years, OCT has become one of the most common imaging technologies used to diagnose and monitor retinal diseases, including AMD. The OCT self-imaging capabilities of the Notal Vision Home OCT (NVHO) system for retinal fluid visualization in the central 10 degrees were validated during several prospective clinical studies1,2,3,4,5. This study is designed to evaluate the retinal fluid exposure of eyes with NV-AMD, using the NVHO system to guide therapy.

DETAILED DESCRIPTION:
Study Design:

This single arm study will enroll up to 15 subjects diagnosed with NV-AMD in at least one eye. Subjects may have previously participated in Notal Home OCT studies. Both eyes of the subjects will be enrolled unless an eye does not meet the inclusion criteria of VA ≥ 20/320. Subjects will be consented and screened. During screening, clinic staff will provide an overview of the NVHO system to subjects. Subjects who meet all screening criteria will be enrolled.

Definitions of the 2 data sources by periods:

Prospective data collected during NVHO guided management period, termed the study period Retrospective data collection during the preceding reference period

Treatment During the Enrollment Visit:

It is expected that enrollment will take place during routine visits, therefore regardless of the fluid status at time of enrollment, it may include standard care anti-VEGF treatment.

Eyes may be enrolled if they were treated recently, and the subject agrees to enroll prior to the next pre-scheduled office visit. The Notal Home OCT system is a non-significant risk investigational device, and it will be used in addition to standard care. NSR letter will be provided to each site.

At Home Setup and Tutorial:

Subjects who meet the inclusion / exclusion criteria will be assigned a NVHO device.

The device will be delivered to the subjects' homes. The subjects will unpack and install the NVHO according to setup guide instructions attached to the package. Upon first usage the subject will undergo an on-device tutorial, explaining how to operate the device and self-image their eyes.

Daily Self-Testing:

Subjects will be instructed to self-image their study eye(s) daily at home for 6 months.

Self-imaging data will be automatically transmitted to the Notal Health Cloud at the end of the daily self-imaging. Volume scans containing 88 B-scans with an average separation of 34 μm over a 3 mm by 3 mm field centered on the fixation point will be generated from the raw scan data for each eye.

Physician Monitoring:

The physician will perform a weekly or frequent review of the NVHO output for all the enrolled eyes from their own study site using an online secured viewer. In addition, the investigator will set a fluid volume notification threshold per fluid type (IRF/SRF/TRF).

The investigator will perform a review within 48 hours from a notification of fluid level reaching the threshold or a time-based review reminder. The details of the flow of the review and corresponding actions are described in the Monitoring Flow Chart Figure 1.

Routine Care / Surveillance Visits:

A routine care visit is planned after 3 months of participation in the study. Following a NVHO review-driven visit, the next routine visit will be rescheduled for 3 months later or will be cancelled if coincides within 4 weeks of the exit visit.

Commercial OCT scan data will be collected during the routine visits. If during a routine visit, the investigator determines that treatment is required, a dedicated treatment visit will be scheduled one week (+/- 2 days) after the routine visit. This is to support office administration and allow the collection of additional data from the NVHO monitoring prior to treatment. The investigators can override the planned schedule at their discretion and document the reason accordingly.

High Frequency Self-Testing Following an Injection:

Following a treatment during the study, the subject will be asked to self-image the study eye every 2-3 hours during daytime hours for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to speak and understand English with fluency. 2. Ability to understand and agree to contents of informed consent either in writing or verbally. 3. At least 55 years of age on date of Screening Visit. 4. Diagnosed with NV-AMD in at least one eye and initiation of anti-VEGF treatment in that eye. 5. Visual Acuity of 20/320 or better. 6. Available and willing to conduct daily self-imaging at home for the duration of the trial.

Exclusion Criteria:

1. Any other retinal disease in the study eye requiring steroidal or anti-VEGF injections (anti-VEGF injections during the study period must be for NV-AMD).
2. Subject's schedule not conducive to completing daily tests at home with the Notal Home OCT device for the duration of the study. -

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include approximately 15 subjects diagnosed with NV-AMD in at least one eye. Subjects may have previously participated in Notal Home OCT studies. Both eyes of the subjects will be enrolled unless an eye does not meet the inclusion criteria of VA ≥20/320. If the eye that does not meet the inclusion criteria is the only eye with NV-AMD, the subject will not be enrolled.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-07-26 (Estimated); Study Completion 2023-09-09 (Estimated)

PRIMARY OUTCOMES:
Area under the fluid volume trajectory between treatments (nl-days) during the study period by fluid type (IRF/SRF/TRF) | 6 months

SECONDARY OUTCOMES:
Percentage of days with successful imaging attempts during daily testing | 6 months
Percentage of days with MSI≥2 and with output eligible for fluid quantification | 6 months
Dates of injections by type of drug during the study period | 6 months
Retina thickness in the central 1 mm circle (CST) and in the entire scan area | 6 months
Area under the fluid volume trajectory between treatments (nl-days) during the reference period by fluid type (IRF/SRF/TRF) | 6 months
Maximal fluid volume reached averaged in a moving window of 3 consecutive testing days during the study period by fluid type (IRF/SRF/TRF) | 6 months
Characteristics of dry AMD (iAMD) eyes converted to NV-AMD and identified with the NVHO, including visual acuity and fluid volume. | 6 months
Time spent by physicians and staff in review of NVHO report and updating the patient's electronic medical record | 6 months
Time spent by physician and staff to communicate with the patients upon enrolment and during scheduling of NVHO related office visits | 6 months
Visual acuity during office visits | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston, Boston, MA.
Locations (3):
- United States (3):
  - Ophthalmic Cons. of Boston, Boston, Massachusetts
  - Pepose Vision Institute, St Louis, Missouri
  - Palmetto Retina Center, Florence, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holekamp NM, de Beus AM, Clark WL, Heier JS. PROSPECTIVE TRIAL OF HOME OPTICAL COHERENCE TOMOGRAPHY-GUIDED MANAGEMENT OF TREATMENT EXPERIENCED NEOVASCULAR AGE-RELATED MACULAR DEGENERATION PATIENTS. Retina. 2024 Oct 1;44(10):1714-1731. doi: 10.1097/IAE.0000000000004167. Epub 2024 Sep 12. PMID 39287534